CLINICAL TRIAL: NCT03127735
Title: An Open-label, Non-randomized, Multicenter Phase I Study to Determine the Maximum Tolerated and / or Recommended Phase II Dose of Oral Mutant IDH1 (mIDH1) Inhibitor BAY1436032 and to Characterize Its Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Clinical Efficacy in Patients With mIDH1-R132X Advanced Acute Myeloid Leukemia (AML)
Brief Title: BAY1436032 in Patients With Mutant IDH1(mIDH1) Advanced Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19036; 2016-004095-22 (EudraCT Number)
Record Dates: First submitted 2017-04-06; First posted 2017-04-25 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Phase 1; mIDH1; IDH1 mutation; mIDH1 inhibitor
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — BAY 1436032

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BAY1436032 (Experimental): Dose escalation:
  Various doses of study drug will be tested on a small number of patients/dose with the goal of identifying the most appropriate dose(s) for further evaluation in dose expansion. The MTD of the study drug may or may not be identified. It is anticipated that 3-4 patients will be treated at each dose of study drug to be tested and that 15-20 total patients will be treated in this part of the trial.
  Dose expansion:
  Up to 2 different doses of study drug will be tested on up to 30 patients/dose with the goal of identifying the most appropriate RP2D for further clinical development. The doses to be evaluated in this part of the trial will be selected based on information obtained during dose escalation.
  Interventions: Drug: BAY1436032

INTERVENTIONS:
Drug: BAY1436032 — BAY1436032 administered continuously as a single agent dosed twice a day orally on Days 1 to 28 of a 28-day cycle.
  Patients may continue treatment with BAY1436032 until disease progression, development of other unacceptable toxicity or Investigator discretion.

SUMMARY:
To determine the maximum tolerated and / or recommended Phase II dose of oral mutant IDH1 (mIDH1) inhibitor BAY1436032 and to characterize its safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary clinical efficacy in patients with mIDH1-R132X advanced acute myeloid leukemia (AML)

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced AML that harbors IDH1 mutation
* Patients are relapsed from or refractory to at least 1 previous line of therapy
* Good kidney and liver function
* Male or female patients
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Women must have a negative serum pregnancy test within 7 days prior to the first dose of study drug or be surgically or biologically sterile or postmenopausal

Exclusion Criteria:

* Previously treated with any prior mIDH1 targeted therapy
* Extramedullary disease only
* History of clinically significant or active cardiac disease
* Active clinically significant infection
* Unresolved chronic toxicity of previous AML treatment
* Taking known strong cytochrome P450 (CYP) 2C8 inducers or inhibitors
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or RP2D of BAY1436032 | Within first 4 weeks of first dose
  If the MTD is not reached during dose escalation, the primary variable will be the recommended phase 2 dose (RP2D) of BAY1436032
Number of participants with Adverse Events as a Measure of | Up to 12 weeks
  As a measure of safety and tolerability

SECONDARY OUTCOMES:
Objective efficacy response | Up to 12 weeks
  Response assessment for AML in this study will be based on the modified Cheson criteria. The following categories are used to capture the investigator's AML response evaluation:
  * Complete remission (CR)
  * Morphologic CR with CRh (morphologic CR with incomplete hematological recovery) and the response category CRp (morphologic CR with incomplete platelet recovery)
  * Partial remission (PR)
  * Response categories for morphologic leukemia-free state (MLFS), stable disease and progressive disease
  * Progressive disease
Duration of response | Up to 12 weeks
  Efficacy data
Event-free survival (EFS) | Up to 12 weeks
  EFS defined as time from start of treatment to treatment failure, relapse, or death due to any cause.
Change of 2 hydroxyglutarate (2-HG) level obtained at baseline and post-baseline | Up to 12 weeks
  Assess pharmacodynamic (PD) effects and evidence of clinical efficacy associated with BAY 1436032 administration in patients. Change from baseline and percent change from baseline will be calculated.
Cmax (maximum observed drug concentration in plasma after a single dose) | Cycle 1 Day 1: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hour post-dose (each cycle is 28 days)
  As a secondary objective of this study evaluate the pharmacokinetics (PK) of BAY 1436032 in patients.
  PK parameters normalized for dose and / or dose and body weight will be calculated.
AUC(0-8) (AUC from time 0 to 8 h after a single dose) | Cycle 1 Day 1: Pre-dose, 0.5, 1, 2, 3, 4, 6, and 8 hour post-dose (each cycle is 28 days)
  As a secondary objective of this study evaluate the pharmacokinetics (PK) of BAY 1436032 in patients.
  PK parameters normalized for dose and / or dose and body weight will be calculated.
AUC(0-12) (AUC from time 0 to 12 h after a single dose) | Cycle 1 Day 1: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hour post-dose (each cycle is 28 days)
  if feasible
Cmax,md (Cmax after multiple doses) | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 12 hour post-dose on Day 15; (each cycle is 28 days)
  As a secondary objective of this study evaluate the pharmacokinetics (PK) of BAY 1436032 in patients.
  PK parameters normalized for dose and / or dose and body weight will be calculated.
AUC(0-8)md (AUC from time 0 to 8 h after multiple doses) | Pre-dose, 0.5, 1, 2, 3, 4, 6, and 8 hour post-dose on Day 15; (each cycle is 28 days)
  As a secondary objective of this study evaluate the pharmacokinetics (PK) of BAY 1436032 in patients.
  PK parameters normalized for dose and / or dose and body weight will be calculated.
AUC(0-12)md (AUC from time 0 to 12 h after multiple doses) | Pre-dose, 0.5, 1, 2, 3, 4, 6, and 8 hour post-dose on Day 15; (each cycle is 28 days)
  if feasible

CONTACTS AND LOCATIONS:
Locations (13):
- United States (8):
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Germany (5):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Medizinische Hochschule Hannover (MHH), Hanover, Lower Saxony
  - Universitätsklinikum Leipzig AöR, Leipzig, Saxony
  - Universitätsklinikum Charite zu Berlin, Berlin
  - Universitätsklinikum Hamburg Eppendorf (UKE), Hamburg